CLINICAL TRIAL: NCT03231553
Title: RCT and Meta-analysis Testing Effectiveness and Cost-effectiveness of a Tailored Text Message Programme (MiQuit) for Smoking Cessation in Pregnancy
Brief Title: Effectiveness and Cost-effectiveness of a Tailored Text Message Programme (MiQuit) for Smoking Cessation in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 17065
Record Dates: First submitted 2017-07-20; First posted 2017-07-27 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Smoking Cessation; Pregnancy Related
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Receive usual NHS antenatal care and any NHS smoking cessation support which they choose to access plus an NHS leaflet giving advice on stopping smoking.
  Receive MiQuit text message cessation programme.
  Interventions: Other: MiQuit text message support programme
- Control (No Intervention): Receive usual NHS antenatal care and any NHS smoking cessation support which they choose to access plus an NHS leaflet giving advice on stopping smoking.

INTERVENTIONS:
Other: MiQuit text message support programme — MiQuit is an automated, responsive text message support programme lasting 12 weeks which sends texts containing self-help smoking cessation support and advice to participants mobile phones.
  Arms: Intervention

SUMMARY:
The trial aims to determine whether or not MiQuit (text-message support programme) is effective when offered in addition to standard behavioural support for smoking cessation in pregnancy.

DETAILED DESCRIPTION:
Smoking in pregnancy is expensive; in the UK in 2010 the annual smoking-attributable maternal and infant health care costs were estimated at up to £87.5 million. In high income countries 13% to 25% of pregnant women smoke and rates are increasing in developing ones. In the UK in 2010 26% of pregnant women smoked with highest rates seen amongst younger, socially disadvantaged women.

However, pregnancy is the life event which most motivates smoking cessation attempts and 50+% of pregnant smokers try stopping, hence smoking cessation support offered in pregnancy is likely to be especially beneficial. Regrettably, in pregnancy, there is only strong efficacy evidence for using either face-to-face or 'self-help' stop smoking support. Although nicotine replacement therapy (NRT) is widely-used by UK pregnant smokers this has at best, borderline efficacy.

Self-help support (SHS) almost doubles the likelihood of smoking cessation in late pregnancy. However SHS programmes which help pregnant smokers to quit were all developed before easily-accessible technologies became widely available.

Text message SHS smoking cessation programmes are highly-acceptable; those trialled with non-pregnant smokers in the US and UK have demonstrated efficacy. Unfortunately, neither programme is appropriate in pregnancy as they make no mention of pregnancy which for most pregnant smokers is the very reason they try quitting; consequently many pregnant smokers would likely find these programmes' advice irrelevant and ignore it.

Funded by CRUK to remedy the lack of acceptable self-help cessation support for pregnant smokers, we developed MiQuit, a text-message, smoking cessation SHS programme for pregnant smokers. MiQuit advice is relevant to pregnancy as it is highly-tailored to gestation. We evaluated MiQuit in two RCTs. The first CRUK-funded trial (n=207) demonstrated acceptability. Subsequently, with NIHR funding we refined MiQuit and tested this in a second RCT which demonstrated the feasibility of recruiting from UK National Health Service (NHS) settings to a multi-centre RCT. Again estimated efficacy was encouraging; in MiQuit and control groups, prolonged abstinence from smoking, validated in late pregnancy was 5.4% and 2.0% respectively.

To efficiently determine whether or not MiQuit works for smoking cessation, we are conducting a third RCT with an almost identical design. The efficacy of the MiQuit system will be assessed by combining the findings, using Trial Sequential Analysis methods, from this trial with the findings from the previous two MiQuit trials. Without requiring an expensive, large RCT this study will tell whether or not MiQuit is efficacious for smoking cessation in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and less than 25 weeks gestation
* Smoking at least 5 cigarettes per day pre-pregnancy
* Smoking at least 1 cigarette on a typical day during pregnancy
* Aged 16 or over
* Agrees to accept information to assist cessation
* Owns or has primary use of a mobile phone
* Familiar with sending and receiving text messages
* Able to understand written English (text messages are in English only) and consent issues explained in English.
* Able to give informed consent

Exclusion Criteria:

* Already enrolled in another text service to assist smoking cessation
* Already enrolled in a smoking cessation study
* Having already participated in the study in an earlier pregnancy

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 1000 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Self-reported abstinence from smoking | 36 weeks gestation
  Self-reported smoking abstinence from 4 weeks after enrolment until 36 weeks gestation, with no more than 5 cigarettes smoked in total between these time points, as reported and biochemically validated at 36 weeks using a cut-point used in the previous two trials.

SECONDARY OUTCOMES:
Self-reported abstinence from smoking at 4 weeks after randomisation | 4 weeks after enrolment
  7 day abstinence reported at 4 weeks
Abstinence from smoking at 36 weeks gestation | 36 weeks gestation
  self-reported and biochemically validated 7 day abstinence at 36 weeks gestation
Use of stop-smoking services | 36 weeks gestation
  use of stop-smoking services
Use of NHS care | At delivery
  Use of NHS care
Birth weight | At delivery
  Weight of infant at birth
Gestational age | At delivery
  Gestational age at birth
Fetal death | At delivery
  Miscarriage or stillbirth
Maternal death | At delivery
  Death of participant
Health Status - baseline | At hospital ante-natal appointment
  Health status measured by EQ-5D-5L at baseline visit
Health Status - 4 weeks after randomisation | 4 weeks post randomisation
  Health status measured by EQ-5D-5L at 4 weeks post randomisation
Health Status - 36 weeks gestation | 36 weeks gestation
  Health status measured by EQ-5D-5L at 36 weeks gestation
Maternal hospital admissions | At delivery
  Hospital admission of participant
Infant hospital admission | At delivery
  Hospital admission of infant
Staff costs | Upto 40 weeks after enrolment
  Overheads and other consumables required to deliver the MiQuit intervention and usual care

CONTACTS AND LOCATIONS:
Overall Officials: Tim Coleman, Study Director — University of Nottingham
Locations (17):
- United Kingdom (17):
  - Royal Berkshire NHS Foundation Trust, Reading, Berkshire
  - Birmingham Womens NHS Foundation Trust, Edgbaston, Birmingham
  - Mid Cheshire Hospitals NHS Trust, Crewe, Cheshire
  - North Cumbria University Hospitals NHS Trust, Carlisle, Cumbria
  - University Hospitals of Derby and Burton NHS Foundation Trust, Derby, Derbyshire
  - Plymouth Hospitals NHS Trust, Plymouth, Devon
  - Pennine Acute Hospitals NHS Trust, Multiple Locations, Greater Manchester
  - East Lancashire Hospitals NHS Trust, Burnley, Lancashire
  - United Lincolnshire Hospitals Trust, Multiple Locations, Lincolnshire
  - Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle, Newcastle Upon Tyne
  - Sherwood Forest Hospitals NHS Trust, Mansfield, Nottinghamshire
  - Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire
  - University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, Staffordshire
  - Northumbria Healthcare NHS Foundation Trust, North Shields, Tyne and Wear
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Countess of Chester Hospital NHS Foundation Trust, Chester
  - City Hospitals Sunderland NHS Foundation Trust, Sunderland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coleman T, Clark M, Welch C, Whitemore R, Leonardi-Bee J, Cooper S, Hewitt C, Jones M, Sutton S, Watson J, Daykin K, Ussher M, Parrott S, Naughton F. Effectiveness of offering tailored text message, self-help smoking cessation support to pregnant women who want information on stopping smoking: MiQuit3 randomised controlled trial and meta-analysis. Addiction. 2022 Apr;117(4):1079-1094. doi: 10.1111/add.15715. Epub 2021 Nov 5. PMID 34636086
- [Derived] Whitemore R, Leonardi-Bee J, Naughton F, Sutton S, Cooper S, Parrott S, Hewitt C, Clark M, Ussher M, Jones M, Torgerson D, Coleman T. Effectiveness and cost-effectiveness of a tailored text-message programme (MiQuit) for smoking cessation in pregnancy: study protocol for a randomised controlled trial (RCT) and meta-analysis. Trials. 2019 May 22;20(1):280. doi: 10.1186/s13063-019-3341-4. PMID 31118090